CLINICAL TRIAL: NCT05617677
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Deucravacitinib in Participants With Active Systemic Lupus Erythematosus (SLE) (POETYK SLE-1)
Brief Title: A Study to Assess Effectiveness and Safety of Deucravacitinib Compared With Placebo in Participants With Active Systemic Lupus Erythematosus (SLE)
Acronym: POETYK SLE-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM011-246; 2022-500699-76 (Other: EU CTR)
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmune Diseases; Immune System Diseases; Connective Tissue Diseases; Immune-mediated Diseases; Active Systemic Lupus Erythematosus; Lupus; SLE; Deucravacitinib; Tyk2; POETYK; POETYK SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Immune System Diseases; Connective Tissue Diseases | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib
- Arm 2: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Arms: Arm 1: Deucravacitinib
Other: Placebo — Specified dose on specified days
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of deucravacitinib compared with placebo in an active moderate to severe Systemic Lupus Erythematosus (SLE) population.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with Systemic Lupus Erythematosus (SLE) at least 24 weeks before the screening visit.
* Meet the European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) 2019 classification criteria for SLE.
* One of the following: positive antinuclear antibodies (ANA) ≥ 1:80 at screening OR positive anti dsDNA OR positive anti Smith (anti Sm) as determined by the central laboratory at screening.
* Total Systemic Lupus Erythematosus Disease Activity Index-2K (SLEDAI-2K) score ≥ 6 points and clinical SLEDAI 2K score ≥ 4 points with joint involvement, and/or cutaneous vasculitis, and/or rash.
* Lupus headache, alopecia, organic brain syndrome, and mucosal ulcers must be recorded on SLEDAI 2K, if indicated, but do not count toward the points required for screening at entry.
* At least one SLE background therapy (immunosuppressant and/or antimalarial) is required for ≥ 12 weeks before the screening visit, must be at a stable dose for ≥ 8 weeks before the screening visit, and must remain stable until randomization and throughout study participation.
* Oral corticosteroid (OCS; prednisone or equivalent) background therapy is permitted but not required. For participants taking OCS, the dose must be stable for ≥ 2 weeks before the screening visit, cannot exceed 30 mg/day at screening, and must remain stable until the Week 4 visit. Participants can be on an OCS as well as an antimalarial and/or an immunosuppressant.

Exclusion Criteria

* Diagnosis of drug-induced SLE rather than idiopathic SLE.
* Other autoimmune diseases (eg, multiple sclerosis, psoriasis, inflammatory bowel disease, etc.) are excluded. Participants with type I autoimmune diabetes mellitus, thyroid autoimmune disease, Celiac disease, or secondary Sjögren's syndrome are not excluded.
* SLE overlap syndromes including, but not limited to, rheumatoid arthritis, scleroderma, and mixed connective tissue disease are excluded.
* Active or unstable lupus neuropsychiatric manifestations, including, but not limited to, any condition defined by BILAG A criteria.
* Active, severe Class III, and IV, lupus nephritis that requires or may require treatment with cytotoxic agents or high-dose CS.
* History of congenital or acquired immunodeficiency.
* Known active infection, or any major episode of infection requiring hospitalization or treatment with parenteral (intramuscular or IV) antimicrobial agents (eg, antibiotics antiviral, antifungal, or antiparasitic agents) within 30 days of randomization, or treatment with oral antimicrobial agents within 2 weeks of randomization.
* Currently on any therapy for chronic infection (eg, pneumocystis, herpes zoster, cytomegalovirus, invasive bacterial or fungal infections, or atypical mycobacteria).
* Taking more than 1 immunosuppressant at screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2028-11-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve Systemic Lupus Erythematosus Responder Index-4 [SRI(4)] response | At week 52

SECONDARY OUTCOMES:
Proportion of participants who achieve British Isles Lupus Assessment Group-based Combined Lupus Assessment (BICLA) response | At week 52
Proportion of participants who achieve both SRI(4) and BICLA (dual responders) | At week 52
Proportion of participants with a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score ≥ 10 at baseline who achieve a CLASI response, defined as a decrease of ≥ 50% from baseline CLASI activity score | At week 52
Proportion of participants who achieve Lupus Low Disease Activity State (LLDAS) | At week 52
Proportion of participants with ≥ 6 active (tender + swollen) joints at baseline who achieve at least 50% from baseline reduction in active (tender + swollen) joints | At week 52
Change from baseline in patient-reported fatigue according to Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue | At week 52
Proportion of participants with oral corticosteroid (OCS) ≥ 7.5 mg/day of prednisone at baseline who are receiving ≤ 5 mg/day of prednisone at Week (Wk) 40 which is maintained through Wk52 and who achieve an SRI(4) response at Wk52. | At Week 52
Number of participants with adverse events (AEs) | Up to 156 weeks
Number of participants with serious adverse events (SAEs) | Up to 156 weeks
Number of participants with AEs leading to discontinuation of treatment | Up to 156 weeks
Number of participants with AEs leading to study discontinuation | Up to 156 weeks
Number of participants with target adverse events of special interest (AESIs) | Up to 156 weeks
Number of participants with laboratory abnormalities | Up to 156 weeks
Number of participants with electrocardiogram (ECG) abnormalities | Up to 156 weeks
Number of participants with vital sign abnormalities | Up to 156 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (197):
- United States (48):
  - Local Institution - 0012, Birmingham, Alabama
  - Local Institution - 0229, Phoenix, Arizona
  - Local Institution - 0193, Tucson, Arizona
  - Kaiser Permanente, Fontana, California
  - Local Institution - 0247, La Mesa, California
  - Local Institution - 0090, La Palma, California
  - Local Institution - 0124, Los Angeles, California
  - Local Institution - 0248, Sacramento, California
  - Local Institution - 0253, San Diego, California
  - Local Institution - 0128, Santa Barbara, California
  - Local Institution - 0099, Denver, Colorado
  - Local Institution - 0054, New Haven, Connecticut
  - Local Institution - 0249, Coral Springs, Florida
  - Local Institution - 0010, Gainesville, Florida
  - Local Institution - 0087, Miami, Florida
  - Local Institution - 0007, Orlando, Florida
  - Local Institution - 0242, Plantation, Florida
  - Local Institution - 0002, Tamarac, Florida
  - Local Institution - 0165, Tampa, Florida
  - Local Institution - 0204, Atlanta, Georgia
  - Local Institution - 0228, Lawrenceville, Georgia
  - Local Institution - 0147, Lawrenceville, Georgia
  - Local Institution - 0227, Morton Grove, Illinois
  - Local Institution - 0077, Schaumburg, Illinois
  - Local Institution - 0108, Indianapolis, Indiana
  - Lake Cumberland Rheumatology, New Albany, Indiana
  - Local Institution - 0225, New Orleans, Louisiana
  - Local Institution - 0006, Detroit, Michigan
  - Local Institution - 0179, Eagan, Minnesota
  - Local Institution - 0177, Summit, New Jersey
  - Local Institution - 0180, Manhasset, New York
  - Local Institution - 0085, New York, New York
  - Local Institution - 0098, Rochester, New York
  - Local Institution - 0159, The Bronx, New York
  - Local Institution - 0245, Charlotte, North Carolina
  - Local Institution - 0155, Charlotte, North Carolina
  - Local Institution - 0246, Summerville, South Carolina
  - Local Institution - 0003, Memphis, Tennessee
  - Local Institution - 0064, Allen, Texas
  - Local Institution - 0065, Dallas, Texas
  - Local Institution - 0088, Fort Worth, Texas
  - Local Institution - 0250, Houston, Texas
  - Local Institution - 0219, Lubbock, Texas
  - Local Institution - 0005, The Woodlands, Texas
  - Local Institution - 0009, Roanoke, Virginia
  - Local Institution - 0011, Seattle, Washington
  - Local Institution - 0139, Seattle, Washington
  - Local Institution - 0063, Franklin, Wisconsin
- Argentina (10):
  - Local Institution - 0078, Quilmes, Buenos Aires
  - Local Institution - 0013, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0020, CABA, Buenos Aires F.D.
  - Local Institution - 0123, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0032, Buenos Aires
  - Local Institution - 0240, Buenos Aires
  - Local Institution - 0022, Buenos Aires
  - Local Institution - 0140, Buenos Aires
  - Local Institution - 0138, Córdoba
  - Local Institution - 0017, Mendoza
- Brazil (12):
  - Local Institution - 0224, Salvador, Estado de Bahia
  - Local Institution - 0096, Lago Sul, Federal District
  - Local Institution - 0042, Belo Horizonte, Minas Gerais
  - Local Institution - 0041, Juiz de Fora, Minas Gerais
  - Local Institution - 0190, Curitiba, Paraná
  - Local Institution - 0181, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0185, Campinas, São Paulo
  - Local Institution - 0187, Ribeirão Preto, São Paulo
  - Local Institution - 0066, São José do Rio Preto, São Paulo
  - Local Institution - 0191, São Paulo, São Paulo
  - Local Institution - 0186, Rio de Janeiro
  - Local Institution - 0125, São Paulo
- Bulgaria (3):
  - Local Institution - 0163, Plovdiv
  - Local Institution - 0217, Sofia
  - Local Institution - 0162, Sofia
- Canada (5):
  - Local Institution - 0126, Calgary, Alberta
  - Local Institution - 0160, Hamilton, Ontario
  - Local Institution - 0114, London, Ontario
  - Local Institution - 0115, Toronto, Ontario
  - Local Institution - 0136, Rimouski, Quebec
- China (32):
  - Local Institution - 0110, Bengbu, Anhui
  - Local Institution - 0070, Beijing, Beijing Municipality
  - Local Institution - 0107, Xiamen, Fujian
  - Local Institution - 0029, Guangzhou, Guangdong
  - Local Institution - 0051, Guangzhou, Guangdong
  - Local Institution - 0080, Guangzhou, Guangdong
  - Local Institution - 0037, Shenzhen, Guangdong
  - Local Institution - 0153, Baoding, Hebei
  - Local Institution - 0133, Luoyang, Henan
  - Local Institution - 0023, Zhengzhou, Henan
  - Local Institution - 0137, Wuhan, Hubei
  - Local Institution - 0044, Changsha, Hunan
  - Local Institution - 0021, Zhuzhou, Hunan
  - Local Institution - 0089, Hohhot, Inner Mongolia
  - Local Institution - 0129, Changzhou, Jiangsu
  - Local Institution - 0031, Jiujiang, Jiangxi
  - Local Institution - 0071, Nanchang, Jiangxi
  - Local Institution - 0117, Nanchang, Jiangxi
  - Local Institution - 0220, Nanchang, Jiangxi
  - Local Institution - 0028, Pingxiang, Jiangxi
  - Local Institution - 0039, Shenyang, Liaoning
  - Local Institution - 0092, Shenyang, Liaoning
  - Local Institution - 0149, Jinan, Shandong
  - Local Institution - 0079, Shanghai, Shanghai Municipality
  - Local Institution - 0045, Shanghai, Shanghai Municipality
  - Local Institution - 0049, Shanghai, Shanghai Municipality
  - Local Institution - 0116, Chengdu, Sichuan
  - Local Institution - 0053, Tianjin, Tianjin Municipality
  - Local Institution - 0043, Ürümqi, Xinjiang
  - Local Institution - 0132, Hangzhou, Zhejiang
  - Local Institution - 0135, Wenzhou, Zhejiang
  - Local Institution - 0158, Taiyuan
- Colombia (7):
  - Local Institution - 0174, Medellín, Antioquia
  - Local Institution - 0056, Barranquilla, Atlántico
  - Local Institution - 0086, Bucaramanga, Santander Department
  - Local Institution - 0100, Bogotá
  - Local Institution - 0170, Bogotá
  - Local Institution - 0093, Cali
  - Local Institution - 0057, Chía
- France (4):
  - Local Institution - 0150, Strasbourg, Alsace
  - Local Institution - 0068, Nantes, Loire-Atlantique
  - Local Institution - 0173, Le Kremlin-Bicêtre
  - Local Institution - 0156, Tours
- Germany (8):
  - Local Institution - 0109, Tübingen, Baden-Wurttemberg
  - Local Institution - 0176, Munich, Bavaria
  - Local Institution - 0146, Dresden, Saxony
  - Local Institution - 0151, Lübeck, Schleswig-Holstein
  - Local Institution - 0195, Chemnitz
  - Local Institution - 0061, Cologne
  - Local Institution - 0120, Erlangen
  - Local Institution - 0111, Planegg
- Local Institution - 0067, Tuenmen, Hong Kong
- India (7):
  - Local Institution - 0213, Vizianagaram, Andhra Pradesh
  - Local Institution - 0200, Ahmedabad, Gujarat
  - Local Institution - 0243, Surat, Gujarat
  - Local Institution - 0208, Gurugram, Haryana
  - Local Institution - 0202, Bengaluru, Karnataka
  - Local Institution - 0222, Hyderabad, Telangana
  - Local Institution - 0205, Hyderabad, Telangana
- Ireland (4):
  - Local Institution - 0119, Manorhamilton, Leitrim
  - Local Institution - 0130, Cork
  - Local Institution - 0157, Dublin
  - Local Institution - 0172, Dublin
- Italy (8):
  - Local Institution - 0084, Rome, Lazio
  - Local Institution - 0095, Milan, Lombardy
  - Local Institution - 0060, Pisa, Tuscany
  - Local Institution - 0097, Padua, Veneto
  - Local Institution - 0069, Brescia
  - Local Institution - 0072, Milan
  - Local Institution - 0154, Napoli
  - Local Institution - 0161, Verona
- Local Institution - 0167, Kaunas, Kaunas County, Lithuania
- Mexico (10):
  - Local Institution - 0015, Mexicali, Estado de Baja California
  - Local Institution - 0082, León, Guanajuato
  - Local Institution - 0024, Zapopan, Jalisco
  - Local Institution - 0026, Mexico City, Mexico City
  - Local Institution - 0027, Mexico City, Mexico City
  - Local Institution - 0016, Mexico City, Mexico City
  - Local Institution - 0050, Mexico City, Mexico City
  - Local Institution - 0112, Mexico City, Mexico City
  - Local Institution - 0018, Chihuahua City
  - Local Institution - 0083, Puebla City
- Moldova (2):
  - Local Institution - 0238, Chisinau, Chișinău
  - Local Institution - 0236, Chisinau
- Peru (4):
  - Local Institution - 0199, Arequipa
  - Local Institution - 0104, Lima
  - Local Institution - 0122, Lima
  - Local Institution - 0103, Lima
- Poland (11):
  - Local Institution - 0036, Poznan, Greater Poland Voivodeship
  - Local Institution - 0040, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0033, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0034, Nadarzyn, Masovian Voivodeship
  - Local Institution - 0164, Warsaw, Masovian Voivodeship
  - Local Institution - 0166, Warsaw, Masovian Voivodeship
  - Local Institution - 0047, Katowice, Silesian Voivodeship
  - Local Institution - 0035, Bialystok
  - Velocity Clinical Research, Lublin, Lublin
  - Local Institution - 0212, Poznan
  - Local Institution - 0211, Bełchatów, Łódź Voivodeship
- Puerto Rico (3):
  - Local Institution - 0203, Caguas
  - Local Institution - 0252, San Juan
  - Local Institution - 0197, San Juan
- Romania (10):
  - Local Institution - 0148, Bucharest, București
  - Local Institution - 0076, Bucharest, București
  - Local Institution - 0152, Bucharest, București
  - Local Institution - 0141, Bucharest, București
  - Local Institution - 0215, Bucharest, București
  - Local Institution - 0210, Bucharest, București
  - Local Institution - 0142, Craiova, Dolj
  - Local Institution - 0216, Iași, Iaşi
  - Local Institution - 0094, Râmnicu Vâlcea, Vâlcea County
  - Local Institution - 0143, Timișoara
- South Korea (4):
  - Local Institution - 0102, Gwangju, Kwangju-Kwangyǒkshi
  - Local Institution - 0101, Suwon, Kyǒnggi-do
  - Local Institution - 0144, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0169, Seoul
- Turkey (Türkiye) (3):
  - Local Institution - 0184, Ankara
  - Local Institution - 0168, Istanbul
  - Local Institution - 0189, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Arriens C, Morand EF, Askanase AD, Furie R, van Vollenhoven RF, Tanaka Y, Connors K, Davey M, Young K, Franchin G, Meier R, Shah V, de Oliveria CL, Hobar C. Design of Two Randomized, Placebo-Controlled, Phase 3 Trials of Deucravacitinib, an Oral, Selective, Allosteric TYK2 Inhibitor, in Systemic Lupus Erythematosus. Adv Ther. 2025 Nov;42(11):5830-5844. doi: 10.1007/s12325-025-03299-0. Epub 2025 Sep 8. PMID 40920289
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05617677.html